CLINICAL TRIAL: NCT01230892
Title: The Evaluation of The Effects of Nebivolol in Comparison to Atenolol on Wall Shear Stress and Rupture Prone Coronary Artery Plaques in Patients With Moderate Coronary Artery Disease
Brief Title: Evaluation of The Effects of Nebivolol in Comparison to Atenolol on Wall Shear Stress and Rupture Prone Coronary Plaques
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Georgia Institute of Technology (Other)
Responsible Party: Principal Investigator, Habib Samady, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00027953; Emory #00000681 (Other: Other)
Record Dates: First submitted 2010-09-10; First posted 2010-10-29 (Estimated); Results first posted 2015-02-27 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Atherosclerosis; Endothelial Function
MeSH Terms: conditions — Atherosclerosis | interventions — Nebivolol; Atenolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nebivolol (Active Comparator)
  Interventions: Drug: Nebivolol
- Atenolol (Active Comparator)
  Interventions: Drug: Atenolol

INTERVENTIONS:
Drug: Nebivolol — 10 mg PO qday
  Other Names: Bystolic
  Arms: Nebivolol
Drug: Atenolol — 100 mg PO qday
  Other Names: Senormin; Tenormin
  Arms: Atenolol

SUMMARY:
Nebivolol is a novel blood pressure lowering drug with an additional effect on the inner lining of blood vessels to release a compound called nitric oxide that can relax blood vessels. Atenolol is a blood pressure reducing agent without the ability to release nitric oxide and effect additional blood vessel relaxation.

The goal of this proposal is to compare Nebivolol and Atenolol with respect to the following parameters:

* Plaque within arteries supplying the heart in terms of its volume and composition as assessed by ultrasound within these arteries.
* Ability of small arteries in the heart to open up and deliver an enhanced blood supply in response to drug called Adenosine (routinely used in the cardiac catheterization laboratory) as assessed by pressure and flow detecting catheters within these arteries.
* Ability of the inner lining of arteries that supply the heart to release a relaxing compound called nitric oxide in response to injection of Acetylcholine (also used in the cardiac catheterization laboratory) as assessed by squirting dye into these arteries
* Local forces that affect blood flow in the arteries supplying the heart as assessed by superimposing the above data into complex maps created offline at Georgia Institute of Technology.

It is likely that Nebivolol causes the plaque within arteries supplying the heart to change from the 'vulnerable' type to the 'stable' type plaque. There are several features of "vulnerable plaques" that can be detected in arteries of the heart using intravascular ultrasound (a small ultrasound camera that goes in the arteries of the heart). The investigators hypothesis is that Nebivolol will prove superior to Atenolol in reducing 'vulnerable plaques', improve blood flow within the small arteries and the health of inner lining of these arteries at the 1 year time point. The investigators plan to enroll 20 patients into the study (26 patient including dropouts) who will be randomized in a 1:1 manner to Nebivolol Vs Atenolol for 1 year and repeat evaluation at that time point.

DETAILED DESCRIPTION:
Primary hypothesis:

Nebivolol therapy will reduce the number of thin-cap fibroatheromas, VH-IVUS defined "vulnerable plaques" compared to Atenolol in patients undergoing serial angiography and IVUS.

Secondary Hypotheses:

* Nebivolol therapy will improve coronary microvascular function
* Nebivolol therapy will improve coronary endothelial function
* Nebivolol therapy will improve coronary wall shear stress

Specific Aims:

To evaluate, in patients with stable angina or acute coronary syndromes and moderate angiographic coronary artery disease, the effects of Nebivolol 5 mg a day compared to Atenolol 50 mg a day on:

* The number of thin cap fibroatheromas, percent necrotic core, and percent atheroma volume as defined by the novel Virtual Histology IVUS (VH™ IVUS).
* The coronary shear stress profile measured using 3 dimensional vessel reconstruction, flow velocity measurements, and computational fluid dynamics.
* Microvascular function as determined by coronary flow reserve and fractional flow reserve measured by invasive Doppler/pressure assessment.
* Endothelial function as determined by the response of quantitative coronary angiography and Doppler assessment to intracoronary acetylcholine challenge.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable angina or acute coronary syndrome
* Moderate coronary lesion (defined as a lesion significant enough by the treating physician to warrant further evaluation using CFR or FFR or intravascular ultrasound assessment).
* Lesion located in the proximal 60mm of the RCA or LAD.
* On stable medical therapy for other cardiac risk factors.

Exclusion Criteria:

* Left Main lesion greater than 50% stenosis
* Patients with a history of coronary artery bypass surgery
* Severe valvular heart disease
* Patients presenting with a STEMI.
* Inability to provide informed consent prior to randomization
* Creatinine >1.5
* Lesions located beyond 60mm in an epicardial vessel
* Coronary anatomy requiring CABG
* B-blocker, calcium channel blocker or extended-release nitrate therapy within last 48 hours.
* Bradycardia (HR<50 bpm)
* Hypotension (SBP<100mmHg)
* Severe COPD by pulmonary function testing

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Habib Samady, MD, FACC, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Hung OY, Molony D, Corban MT, Rasoul-Arzrumly E, Maynard C, Eshtehardi P, Dhawan S, Timmins LH, Piccinelli M, Ahn SG, Gogas BD, McDaniel MC, Quyyumi AA, Giddens DP, Samady H. Comprehensive Assessment of Coronary Plaque Progression With Advanced Intravascular Imaging, Physiological Measures, and Wall Shear Stress: A Pilot Double-Blinded Randomized Controlled Clinical Trial of Nebivolol Versus Atenolol in Nonobstructive Coronary Artery Disease. J Am Heart Assoc. 2016 Jan 25;5(1):e002764. doi: 10.1161/JAHA.115.002764. PMID 26811165

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nebivolol | Atenolol
Started | 15 | 14
Completed | 12 | 13
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Population: 4 subjects either withdrew or were lost to follow-up and not included in analysis population. Additionally, one subject in the Atenolol arm was removed from analysis population due to IVUS occurring in the incorrect artery.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebivolol | Atenolol | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (10) | 50 (11) | 52 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 8 | 10 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reduction of Thin-cap Fibroatheromas (TCFA) as Defined by VH-IVUS
Description: Presence of thin-cap fibroatheroma as defined by virtual histology-intravascular ultrasound (VH-IVUS)
Time Frame: 1 year
Population: 4 subjects either withdrew or were lost to follow-up and not included in analysis population. Additionally, one subject in the Atenolol arm was removed from analysis population due to IVUS occurring in the incorrect artery and one subject in the Nebivolol arm was removed due to the IVUS catheter malfunctioning.
Measure: Number; unit: participants
Arm/Group | Nebivolol | Atenolol
Number analyzed (Participants) | 11 | 12
participants | 4 | 6

ADVERSE EVENTS:
Arm/Group | Nebivolol | Atenolol
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 0/15 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No